CLINICAL TRIAL: NCT01879384
Title: Feasibility of Monitoring of Bone Free Flaps With Microdialysis Catheter Directly Positioned in Bone Tissue
Brief Title: Monitoring of Bone Free Flaps With Microdialysis
Acronym: MTM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Collaborators: Regional Council Picardie (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PI08-PR-DEVAUCHELLE; 2010-A01176-33 (Other: ID-RCB)
Record Dates: First submitted 2013-06-13; First posted 2013-06-17 (Estimated); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Microsurgery; Head and Neck Reconstructive Surgery; Head and Neck Cancer; Head and/or Neck Shotgun Trauma; Bone Free Flap
Keywords: microdialysis; bone free flap; head and neck; monitoring free flap; reconstructive surgery
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Microdialysis with CMA 70 catheter (Experimental): CMA 70 catheter directly positioned in bone tissue
  Interventions: Device: CMA 70 catheter directly positioned in bone tissue

INTERVENTIONS:
Device: CMA 70 catheter directly positioned in bone tissue — At the end of the surgery the CMA microdialysis catheter is placed inside the bone

SUMMARY:
Microdialysis is admitted to be reliable by numerous surgeons to monitor flaps. Nevertheless, a few authors reported follow up with microdialysis in bone flaps, and they all described the position of the catheter in the surrounding soft tissue muscle. This surrounding soft tissue is not always the reflect of bone vascularisation.

The aim is to study the feasibility of a follow up of microanastomosed bone flaps with microdialysis. To reach this goal, investigators perform a clinical prospective research project untitled MTM project

DETAILED DESCRIPTION:
In addition to our classical clinical monitoring, bone microanastomosed flaps for reconstructive facial surgery will be monitored with CMA 70 catheter directly positioned in bone tissue.

The monitoring is recorded during 5 days. Glucose, lactate , pyruvate , glycerol rates will be analysed :

* every hour at day 1,
* every two hours at day 2,
* every three hours at day 3,4 and 5.

Data are managed with Labpilot software.

ELIGIBILITY:
Inclusion Criteria:

* head and neck reconstruction with iliac crest or fibula free flaps
* informed consent obtained

Exclusion Criteria:

* reconstruction with other types of free flaps

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2011-02; Primary Completion 2013-05 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Feasibility study of monitoring bone free flaps with microdialysis (catheter directly positioned in bone tissue) | Day 5 after catheter insertion
  Success of microdialysis is defined as the collection and measurement of metabolites levels as: lactate, pyruvate,glycerol and glucose.

SECONDARY OUTCOMES:
Evaluation of "flush-out" period | Day 5 after catheter insertion
  Time required to acquire interpretable data after opening microdialysis circuit
Compliance of the prescription | Day 5 after catheter insertion
  Compliance rate of simples collected and analysed

OTHER OUTCOMES:
Delay of ischemia detection with metabolic parameters, compared to clinical symptoms | from implantation time day 5
  Time between the occurrence of the first metabolic changes and the first clinical signs of tissue damage

CONTACTS AND LOCATIONS:
Overall Officials: Bernard DEVAUCHELLE, MD, phD, Principal Investigator — Amiens University Hospital
Locations (1):
- Amiens University Hospital, Amiens, Picardie, France

REFERENCES:
- [Background] Abdel-Galil K, Mitchell D. Postoperative monitoring of microsurgical free-tissue transfers for head and neck reconstruction: a systematic review of current techniques--part II. Invasive techniques. Br J Oral Maxillofac Surg. 2009 Sep;47(6):438-42. doi: 10.1016/j.bjoms.2008.12.002. Epub 2009 Jan 19. PMID 19155107
- [Background] Benacquista T, Kasabian AK, Karp NS. The fate of lower extremities with failed free flaps. Plast Reconstr Surg. 1996 Oct;98(5):834-40; discussion 841-2. doi: 10.1097/00006534-199610000-00013. PMID 8823023
- [Background] Birke-Sorensen H, Toft G, Bengaard J. Pure muscle transfers can be monitored by use of microdialysis. J Reconstr Microsurg. 2010 Nov;26(9):623-30. doi: 10.1055/s-0030-1267382. Epub 2010 Oct 6. PMID 20927696
- [Background] Bogehoj M, Emmeluth C, Overgaard S. Blood flow and microdialysis in the human femoral head. Acta Orthop. 2007 Feb;78(1):56-62. doi: 10.1080/17453670610013420. PMID 17453393
- [Background] Brix M, Muret P, Ricbourg B, Humbert P. [Monitoring free flaps with cutaneous microdialysis: preliminary study in oral cavity reconstruction]. Rev Stomatol Chir Maxillofac. 2006 Dec;107(6):460-4. doi: 10.1016/s0035-1768(06)77088-7. French. PMID 17195000
- [Background] Bui DT, Cordeiro PG, Hu QY, Disa JJ, Pusic A, Mehrara BJ. Free flap reexploration: indications, treatment, and outcomes in 1193 free flaps. Plast Reconstr Surg. 2007 Jun;119(7):2092-2100. doi: 10.1097/01.prs.0000260598.24376.e1. PMID 17519706
- [Background] Delgado JM, DeFeudis FV, Roth RH, Ryugo DK, Mitruka BM. Dialytrode for long term intracerebral perfusion in awake monkeys. Arch Int Pharmacodyn Ther. 1972;198(1):9-21. No abstract available. PMID 4626478
- [Background] Ferguson REH Jr, Yu P. Techniques of monitoring buried fasciocutaneous free flaps. Plast Reconstr Surg. 2009 Feb;123(2):525-532. doi: 10.1097/PRS.0b013e318196b9a3. PMID 19182610
- [Background] Holzle F, Rau A, Loeffelbein DJ, Mucke T, Kesting MR, Wolff KD. Results of monitoring fasciocutaneous, myocutaneous, osteocutaneous and perforator flaps: 4-year experience with 166 cases. Int J Oral Maxillofac Surg. 2010 Jan;39(1):21-8. doi: 10.1016/j.ijom.2009.10.012. Epub 2009 Nov 26. PMID 19944567
- [Background] Jallali N, Ridha H, Butler PE. Postoperative monitoring of free flaps in UK plastic surgery units. Microsurgery. 2005;25(6):469-72. doi: 10.1002/micr.20148. PMID 16134095
- [Background] Jyranki J, Suominen S, Vuola J, Back L. Microdialysis in clinical practice: monitoring intraoral free flaps. Ann Plast Surg. 2006 Apr;56(4):387-93. doi: 10.1097/01.sap.0000205231.39853.87. PMID 16557069
- [Background] Laure B, Sury F, Bayol JC, Goga D. [Microdialysis: experience in postoperative monitoring of 30 free flaps]. Ann Chir Plast Esthet. 2009 Feb;54(1):29-36. doi: 10.1016/j.anplas.2008.05.008. Epub 2008 Nov 29. French. PMID 19042067
- [Background] Mourouzis C, Anand R, Bowden JR, Brennan PA. Microdialysis: use in the assessment of a buried bone-only fibular free flap. Plast Reconstr Surg. 2007 Oct;120(5):1363-1366. doi: 10.1097/01.prs.0000279555.75241.4c. No abstract available. PMID 17898613
- [Background] Rojdmark J, Blomqvist L, Malm M, Adams-Ray B, Ungerstedt U. Metabolism in myocutaneous flaps studied by in situ microdialysis. Scand J Plast Reconstr Surg Hand Surg. 1998 Mar;32(1):27-34. doi: 10.1080/02844319850158921. PMID 9556818
- [Background] Setala L, Papp A, Romppanen EL, Mustonen P, Berg L, Harma M. Microdialysis detects postoperative perfusion failure in microvascular flaps. J Reconstr Microsurg. 2006 Feb;22(2):87-96. doi: 10.1055/s-2006-932502. PMID 16456768
- [Background] Setala LP, Korvenoja EM, Harma MA, Alhava EM, Uusaro AV, Tenhunen JJ. Glucose, lactate, and pyruvate response in an experimental model of microvascular flap ischemia and reperfusion: a microdialysis study. Microsurgery. 2004;24(3):223-31. doi: 10.1002/micr.20045. PMID 15160382
- [Background] Smit JM, Zeebregts CJ, Acosta R, Werker PMN. Advancements in free flap monitoring in the last decade: a critical review. Plast Reconstr Surg. 2010 Jan;125(1):177-185. doi: 10.1097/PRS.0b013e3181c49580. PMID 20048610
- [Background] Stolle LB, Arpi M, Jorgensen PH, Riegels-Nielsen P, Keller J. In situ gentamicin concentrations in cortical bone: an experimental study using microdialysis in bone. Acta Orthop Scand. 2003 Oct;74(5):611-6. doi: 10.1080/00016470310018045. PMID 14620985
- [Background] Ungerstedt U, Rostami E. Microdialysis in neurointensive care. Curr Pharm Des. 2004;10(18):2145-52. doi: 10.2174/1381612043384105. PMID 15281890
- [Result] Dakpe S, Colin E, Bettoni J, Davrou J, Diouf M, Devauchelle B, Testelin S. Intraosseous microdialysis for bone free flap monitoring in head and neck reconstructive surgery: A prospective pilot study. Microsurgery. 2020 Mar;40(3):315-323. doi: 10.1002/micr.30529. Epub 2019 Oct 22. PMID 31638286